CLINICAL TRIAL: NCT02504996
Title: IV Paracetamol vs IV Morphine vs Placebo in Sciatalgia in Patients Presented With Sciatalgia to Emergency Department: A Randomized Controlled Trial
Brief Title: IV Paracetamol vs IV Morphine vs Placebo in Sciatalgia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Collaborators: Pamukkale University (Other); Antalya Training and Research Hospital (Other Government); University of Gaziantep (Other); Ataturk University (Other)
Responsible Party: Principal Investigator, Cenker Eken, Associate Proffesor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 70178
Record Dates: First submitted 2015-07-02; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Sciatica
Keywords: sciatalgia; emergency department; paracetamol; morphine
MeSH Terms: conditions — Sciatica; Emergencies | interventions — Acetaminophen; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Paracetamol (Active Comparator): 1 g intravenous paracetamol (Perfalga, Bristol Myers) in 100 ml saline with a rapid infusion.
  Interventions: Drug: Paracetamol
- morphine (Active Comparator): 0.1 mg/kg morphine in 100 ml saline with a rapid infusion.
  Interventions: Drug: morphine
- placebo (Placebo Comparator): 100 ml saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol — 1 g paracetamol via intravenous route in 100 ml normal saline
  Other Names: Perfalgan
  Arms: Paracetamol
Drug: morphine — 0.1 mg/kg morphine via intravenous route in 100 ml normal saline
  Other Names: Morfin
  Arms: morphine
Drug: Placebo — Intravenous 100 ml normal saline
  Arms: placebo

SUMMARY:
Siatalgia is one of the main symptoms related to emergency department presentations. Patients with sciatalgia are seeking for immediate pain relief and little known regarding the pain management of these patients in emergency department. This study aim to trial the effect of intravenous paracetamol and morphine in patients presented with sciatalgia to emergency department.

DETAILED DESCRIPTION:
Siatalgia is one of the main symptoms related to emergency department presentations. Patients with sciatalgia are seeking for immediate pain relief and little known regarding the pain management of these patients in emergency department. Neuronal compression is the main cause of pain in sciatalgia rather than inflammation which also differ sciatalgia from the other type of pains in emergency department. Sciatalgia is a kind of neuralgia and there is not so much option in the pain management of these patients. Intravenous paracetamol and morphine is commonly used analgesics in various kind of pain in emergency department. So, this study aim to trial the effect of intravenous paracetamol and morphine in patients presented with sciatalgia to emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pain radiating to the sciatic nerve path
* Pain within the last one week
* Patients with positive straight leg raise
* Patients over 21 and lower than 65 years old

Exclusion Criteria:

* Pain score lower than 40 mm in visual analogue scale score
* Neurological deficit
* Allergy to the study drugs
* Unstable vital signs
* History of malignancy or rheumatological diseases or arthritis
* History of chronic pain syndrome
* Receiving pain killer, steroid, anti-depressant, anti-convulsant and musculorelaxant within the last six hours.
* Drug or alcohol addiction
* Pregnancy or breast feeding
* Fewer more than 37.9 Celsius degrees.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale Score to measure pain reduction | 30 minutes
  Visual Analogue Scale Score at 30 minutes in order to measure pain reduction

SECONDARY OUTCOMES:
Rescue drug need questionnaire | 30 minutes
  The rescue drug need will be recorded by asking the study patient at 30 minutes. yes/no
Adverse effects | 30 minutes
  Adverse effects occurred within the 30 minutes period

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Serinken, MD, Study Chair — Pamukkale University
Locations (1):
- Pamukkale University Hospital, Denizli, Turkey (Türkiye)